CLINICAL TRIAL: NCT00147550
Title: A Multicenter, Open-Label, Noncomparative Phase 1-2 Clinical And Pharmacokinetic Study Of Oral PD 0325901 In Patients With Advanced Cancer
Brief Title: MEK Inhibitor PD-325901 To Treat Advanced Breast Cancer, Colon Cancer, And Melanoma.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4581001
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2013-09

CONDITIONS: Melanoma; Colonic Neoplasms; Breast Neoplasms
MeSH Terms: conditions — Melanoma; Colonic Neoplasms; Breast Neoplasms | interventions — mirdametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: PD-0325901

INTERVENTIONS:
Drug: PD-0325901 — Administered orally either once or twice a day; several dosing schedules evaluated; current dosing schedule is 5 days on-drug, 2-days off drug for 3 weeks in a 28-day cycle. Doses evaluated ranged from 1 mg once a day to 30 mg twice daily.

SUMMARY:
MEK is a critical member of the MAPK pathway involved in growth and survival of cancer cells. PD-325901 is a new drug designed to block this pathway and kill cancer cells. The purpose of this study is to study the effectiveness of PD-325901 in patients with colon cancer, breast cancer, and melanoma. PD-325901 will be given by mouth as a pill twice a day, CT scans will be done and biopsies will be taken of a tumor before and once during treatment to measure the effects of the drug. Blood samples will be taken to measure the amount of drug in the blood.

DETAILED DESCRIPTION:
The study prematurely discontinued on March 15, 2007 due to a safety concern, specifically ocular and neurological toxicity presented at 10 mg twice-a-day and higher doses.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years old
* Tumor accessible for biopsy and willingness to undergo baseline and 1 post treatment biopsy
* Biopsiable, histologically or cytologically confirmed metastatic or inoperable breast cancer, colon cancer, or melanoma. Prior treatment requirement : i) no more than 2 prior cytotoxic chemotherapy regimens for metastatic disease for patients with breast or colon cancers; ii) No prio cytotoxic therapy for patients with melanoma, or iii) measurable lesion (s) that have not been irradiated.
* Adequate renal, liver, and bone marrow function, determined within 2 weeks prior to the first treatment, defined as the following: Serum creatinine <1.5 x ULN, total bilirubin <2 x ULN, aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <3 x ULN (<5 x ULN for patients with liver involvement); absolute neutrophil count (ANC) >1500/ul; and platelet >100,000/ul
* Hemoglobin >9.0 g/dL. Treatment with transfusions or erythropoietin to elevate the hemoglobin level for eligibility purposes is not permitted. Patients must have discontinued erythropoietin at least 2 weeks prior to the first dose of study medication
* Serum calcium <1 x ULN and phosphorus <1 x ULN
* Patients having reproductive potential must use adequate method of birth control. Patients may not be pregnant or breastfeeding.
* ECOG Status of 0,1, or 2.
* Must be able to swallow intact study medication and have no gastrointestinal disorders that may affect absorption of the drug
* Must be able to follow instructions or protocol specified procedures, or have a daily care giver who will be responsible for administering study medication.
* Must be able to give written informed consent.

Exclusion Criteria:

* No parathyroid disorder or history of malignancy associated hypercalcemia
* No ongoing radiation therapy or radio-cytotoxic therapy within prior 4 weeks; No immunotherapy, biologic therapy, hormonal, or molecular targeted therapy within prior 2 weeks
* No concurrent serious infection or life-threatening illness (unrelated to tumor)
* No history of any cancer other than the present condition (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 3 years
* No untreated brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2004-02; Primary Completion 2007-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate, Safety. | duration of trial

SECONDARY OUTCOMES:
Time to progression, overall survival, patient reported outcomes. | duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, La Mesa, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Santa Monica, California
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Detroit, Michigan
  - Pfizer Investigational Site, Rochester, Minnesota
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Cleveland, Ohio

REFERENCES:
- [Derived] Boasberg PD, Redfern CH, Daniels GA, Bodkin D, Garrett CR, Ricart AD. Pilot study of PD-0325901 in previously treated patients with advanced melanoma, breast cancer, and colon cancer. Cancer Chemother Pharmacol. 2011 Aug;68(2):547-52. doi: 10.1007/s00280-011-1620-1. Epub 2011 Apr 24. PMID 21516509
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4581001&StudyName=MEK%20Inhibitor%20PD-325901%20To%20Treat%20Advanced%20Breast%20Cancer%2C%20Colon%20Cancer%2C%20And%20Melanoma.